CLINICAL TRIAL: NCT05200494
Title: Assessment of Lung Aeretion After Flexible Bronchoscopy for Secretion Removal in Intubated Critically Ill Patients Receiving or Not a Recruiting Maneuver Soon After the Procedure: an Observational Physiological Study
Brief Title: Lung Aeration After Flexible Bronchoscopy in Intubated Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ICU Bronchoscopy
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Failure
Keywords: Secretions; Bronchoscopy; Lung Ultrasound; Electrical Impedance Tomography

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive or not a Recruiting Maneuver (RM) at the end of the Flexible Bronchoscopy. RM will be performed by the application to the airways of 30 cmH2O positive pressure for 30 seconds.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked since he/she will be not present at the end of the procedure, when the intervention (Recruiting Maneuver) will be applied or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Bronchoscopy without Recruiting Maneuver (No Intervention): At the end of the bronchoscopy, no further interventions or ventilator maneuvers will be done.
- Flexible Bronchoscopy with Recruiting Maneuver (Experimental): At the end of the bronchoscopy, a recruiting maneuver will be applied to the patients. Recruiting Maneuver consists in the application of an airway pressure of 30 cmH2O for a period of 30 seconds.
  Interventions: Procedure: Recruiting Maneuver

INTERVENTIONS:
Procedure: Recruiting Maneuver — Airway pressure will be increased to 30 cmH2O for 30 seconds at the end of the bronchoscopy
  Arms: Flexible Bronchoscopy with Recruiting Maneuver

SUMMARY:
In patients suffering from acute respiratory failure, ineffective cough and the consequent retention of secretions are common clinical problems, which often lead to the need for tracheostomy for the sole purpose of aspiration of secretions from the airways.

Mechanically ventilated critically ill patients often have impaired mucus transport which is associated with secretion retention and subsequent development of pneumonia. The accumulation of tracheobronchial secretions in ventilated patients in ICU is due not only to an increased production, but also to a decreased clearance. In the event that secretions occlude a bronchus, an atelectasis of the lung parenchyma is created downstream. Therefore, it is often necessary to perform a flexible bronchoscopy (FOB) to proceed with the removal of the secretion plug. After its removal, the lung is supposed to be reventilated and recruited.

In intubated ICU patients, the application of a recruiting maneuver (RM) is commonly used to reopen the collapsed lung in patients with Acute Respiratory Distress Syndrome or in case of atelectasis in other clinical conditions. However, no studies have so far investigated the role of the application of a RM after a FOB performed to remove a secretion plug in intubated ICU patients.

This observational and physiological study aims to assess if the application of a RM would modify the lung aeration soon after an FOB to remove secretion plug (first outcome). Moreover, the study aims to assess if EIT could be an additional bedside imaging tool to monitor modifications of lung ventilation and aeration during and after a flexible bronchoscopy, as compared with both chest-X-ray and lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation
* need for flexible bronchoscopy to remove secretion plug from the airway

Exclusion Criteria:

* hemodynamic instability, (i.e. systolic arterial pressure <90 mmHg or mean systolic pressure <65 mmHg despite fluid repletion);
* need for vasoactive agents, i.e. vasopressin or epinephrine at any dosage, or norepinephrine >0.3 mcg/kg/min or dobutamine>5 mcg/kg/min;
* life-threatening arrhythmias or electrocardiographic signs of ischemia;
* contraindications to placement of Electrical Impedance Tomography belt, Lung UltraSound or application of a Recruiting Maneuver (i.e., pneumothorax, pulmonary emphysema, chest burns or thoracic surgery within 1 week);
* inclusion in other research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung Aeration through EIT | One hour after the end of the bronchoscopy
  Improvement of lung aeration will be assess with End Expiratory Lung Impedance through Electrical Impedance Tomography, as compared to baseline (before the bronchoscopy)
Lung Aeration through Lung Ultrasound | One hour after the end of the bronchoscopy
  Improvement of lung aeration will be assess with Lung Ultrasound Score, as compared to baseline (before the bronchoscopy)

SECONDARY OUTCOMES:
Arterial Blood Gases | Soon after the end of the bronchoscopy
  Arterial Blood Gases will be assessed through an arterial blood sample
Arterial Blood Gases | One hour after the end of the bronchoscopy
  Arterial Blood Gases will be assessed through an arterial blood sample
Lung Aeration through EIT | Soon after the end of the bronchoscopy
  Improvement of lung aeration will be assess with End Expiratory Lung Impedance through Electrical Impedance Tomography, as compared to baseline (before the bronchoscopy)
Lung Aeration through Lung Ultrasound | Soon after the end of the bronchoscopy
  Improvement of lung aeration will be assess with Lung Ultrasound Score , as compared to baseline (before the bronchoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared after study publication on a peer-reviewed journal in english language, on a reasonable request to the principal investigator
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After study publication on a peer-reviewed journal in english language
Access Criteria: On reasonable request to the Principal Investigator